CLINICAL TRIAL: NCT04084457
Title: Randomised, Double-blind, Placebo Controlled, Parallel Trial Investigating the Daily Effects of Blueberry (Poly)Phenol Consumption on Vascular Function and Cognitive Performance in Healthy Elderly Individuals
Brief Title: Investigating the Effects of Daily Consumption of Blueberry (Poly)Phenols on Vascular Function and Cognitive Performance
Acronym: BluFlow
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: University of Reading (Other)
Responsible Party: Principal Investigator, Dr Ana Rodriguez-Mateos, Principal Investigator, King's College London
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BluFlow
Record Dates: First submitted 2019-09-02; First posted 2019-09-10 (Actual); Last update posted 2021-07-12 (Actual); Status verified 2021-07

CONDITIONS: Healthy Aging; Healthy
Keywords: polyphenols; Blueberries; cognition; vascular function; vascular health; cognitive function; anthocyanins; flavonoids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Matched for macronutrients, micronutrients and fibre
  Interventions: Dietary Supplement: Placebo
- Wild Blueberry Powder (Active Comparator): Formulation of a 100% blueberry (freeze-dried whole fruit) drink
  Interventions: Dietary Supplement: Wild Blueberry powder

INTERVENTIONS:
Dietary Supplement: Wild Blueberry powder — Powdered extract obtained from wild blueberries. A daily administration of 27g wild blueberry powder will be administered.
  Arms: Wild Blueberry Powder
Dietary Supplement: Placebo — Identical formulation as the treatment matched for fibre and vitamin C
  Arms: Placebo

SUMMARY:
Foods rich in certain (poly)phenols, particularly flavonoids, such as berries and cocoa, have been shown to improve measures of vascular function as well as cognitive performance in human intervention studies. This is a randomized, double-blind, placebo controlled, parallel trial investigating the effects of daily blueberry (poly)phenol consumption on vascular function and cognitive performance in healthy elderly individuals. The study will be conducted at King's College London, Franklin-Wilkins Building.

Eligible subjects will be healthy males and females aged 65-80.

DETAILED DESCRIPTION:
To date no study has investigated whether daily blueberry consumption can induce an increase in cerebral blood flow, with subsequent improvements in vascular and cognitive function. In this study, the investigators aim to directly link daily blueberry consumption with improved vascular function, increased cerebral blood flow and positive cognitive outcomes in healthy elderly individuals. The investigators will use a large group of elderly individuals' representative of a healthy population, both males and females, aged 65-80 years to evaluate the health effects of daily blueberry consumption.

The main aim is to investigate whether improvements in vascular and cognitive function previously seen after blueberry consumption can be seen following 3-months daily consumption in elderly individuals, and whether enhanced cognitive performance is correlated with increased cerebral blood flow. The investigators hypothesise that daily consumption of an anthocyanin rich blueberry drink will improve cognitive performance and vascular function, increasing cerebral blood flow, in healthy older individuals.

ELIGIBILITY:
Inclusion Criteria:

* Participants will include 60 healthy male and female volunteers, aged 65-80.
* Volunteers will be able to understand the nature of the study and able to give signed written informed consent.
* Subjects willing to maintain their normal eating/drinking habits and exercise habits to avoid changes in body weight over the duration of the study.

Exclusion Criteria:

* Manifest cardiovascular diseases including coronary artery disease, cerebrovascular disease and peripheral artery disease.
* Hypertensive, as defined as SBP superior or equal to 140 mmHg or DBP superior or equal to 90 mmHg.
* Obese participants, defined as BMI superior or equal to 30.
* Diabetes mellitus and metabolic syndrome.
* Acute inflammation, terminal renal failure or malignancies.
* Allergies to berries or another significant food allergy.
* Subjects under medication or on vitamin/dietary supplements (within 2 weeks of baseline).
* Subjects who have lost more than 10% of their weight in the past 6 months or are currently on a diet.
* Subjects who reported participant in another study within one month before the study starts.
* Subjects who smoke cigarettes irregularly.
* MCI or dyslexic or unable to complete the cognitive function tasks for any reason such as visual impairments.
* Subjects who require chronic antimicrobial or antiviral treatment.
* Subjects with unstable psychological condition.
* Subjects with history of cancer, myocardial infarction, cerebrovascular incident.
* Any reason or condition that in the judgment of the clinical investigator(s) may put the subject at unacceptable risk or that may preclude the subject from understanding or complying with the study's requirements.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-04-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Endothelial Function | Baseline and 12 weeks post-intervention
  Changes in flow-mediated dilation of the brachial artery (FMD) from baseline after 12-week consumption of blueberry vs control
Cognitive function | Baseline and 12 weeks post-intervention
  Changes in cognitive function from baseline after 12-week consumption of blueberry vs control. Cognitive testing involves the participant conducting tasks administered on a tablet-style laptop. The participants will be conducting these tasks whilst cerebral blood flow measurements are taking place. The cognitive testing battery will consist of 4 tasks which are Auditory Verbal learning task, Corsi Blocks, Switching task and Serials 3's and 7's, including a mood assessment (PANAS).

SECONDARY OUTCOMES:
Cerebral blood flow velocity (CBFv) | Baseline and 12 weeks post-intervention
  Changes in cerebral blood flow velocity (CBFv) from baseline after 12-week consumption of blueberry vs control. Trans-cranial blood flow will be assessed by Non-imaging transcranial Doppler sonography (TCD). Variables measured include resting and active mean blood flow velocity (cm/s).
Office systolic blood pressure | Baseline and 12 weeks post-intervention
  Changes from baseline office systolic blood pressure (mmHg) after 12-week consumption of blueberry vs control.
Pulse wave velocity (PWV) | Baseline and 12 weeks post-intervention
  Determine the changes in Pulse wave velocity (PWV) from baseline after 12-week consumption of blueberry vs control.
Augmentation Index (AIx) | Baseline and 12 weeks post-intervention
  Changes in augmentation Index (AIx) using a Sphygmocor device post consumption of a placebo or blueberry treatment
24-hour ambulatory systolic blood pressure | Baseline and 12 weeks post-intervention
  Determine the effect of the blueberry extract vs Placebo on 24-hour systolic blood pressure using a monitor, at 12 weeks post consumption. Variables include mean asleep, awake and total 24 h systolic blood pressure
Mood | Baseline and 12 weeks post-intervention
  Assessment using a self-reported questionnaire using the Positive and Negative Affect Schedule (PANAS).PANAS (The Positive and Negative Affect Schedule) to measure mood, where the participants will need to answer 20 questions using a 5-point likert scale that ranges from (1) not at all to (5) extremely. Dependent variables are composite positive affect and negative affect scores obtained by summing responses to positive or negative PANAS items, respectively.
Change in Blood lipids concentration (Total, HDL and LDL cholesterol, triglycerides) | Baseline and 12 weeks post-intervention
  Determine the effect of the blueberry extract vs Placebo on blood lipids (Total, HDL and LDL cholesterol, triglycerides), at 12 weeks post consumption.
Plasma blueberry (poly)phenol metabolites | Baseline and 12 weeks post-intervention
  Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours post consumption
Microbiome analysis | Baseline and 12 weeks post-intervention
  Stool sample collection involving an all-in-one kit for self-collection and stabilization of microbial DNA from faeces for gut microbiome profiling.
Urine blueberry polyphenol metabolites | Baseline and 12 weeks post-intervention
  Collected over a 24 hour period. Measured by liquid chromotography- mass spectrometry (LC/MS) 0 and 2 hours post consumption
Number of volunteers with treatment-related adverse events | Baseline and 12 weeks post-intervention
  The number of volunteers with treatment-related adverse events will be assessed by questionnaires and interviews.
Pulsatility index (PI) | Baseline and 12 weeks post-intervention
  Changes in pulsatility index (PI) from baseline after 12-week consumption of blueberry vs control. Trans-cranial blood flow will be assessed by Non-imaging transcranial Doppler sonography (TCD). Variables measured include resting and active PI (cm/s.
Office diastolic blood pressure | Baseline and 12 weeks post-intervention
  Changes from baseline office diastolic blood pressure (mmHg) after 12-week consumption of blueberry vs control.
24-hour ambulatory diastolic blood pressure | Baseline and 12 weeks post-intervention
  Determine the effect of the blueberry extract vs Placebo on 24-hour diastolic blood pressure using a monitor, at 12 weeks post consumption. Variables include mean asleep, awake and total 24 h diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Ana Rodriguez-Mateos, PhD, Principal Investigator — Principal Investigator
Locations (1):
- Franklin-Wilkins Building, King's College London, London, United Kingdom

REFERENCES:
- [Derived] Wood E, Hein S, Mesnage R, Fernandes F, Abhayaratne N, Xu Y, Zhang Z, Bell L, Williams C, Rodriguez-Mateos A. Wild blueberry (poly)phenols can improve vascular function and cognitive performance in healthy older individuals: a double-blind randomized controlled trial. Am J Clin Nutr. 2023 Jun;117(6):1306-1319. doi: 10.1016/j.ajcnut.2023.03.017. Epub 2023 Mar 25. PMID 36972800